CLINICAL TRIAL: NCT05685680
Title: Outcome of Laparoscopic Total Mesorectal Excision Versus Open Technique in Management of Rectal Carcinoma
Brief Title: Outcome of Laparoscopic Total Mesorectal Excision Versus Open Technique in Management of Rectal Carcimoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Osama Saleh Ahmed, Assistant lecture ofgeneral surgery, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-12-17
Record Dates: First submitted 2022-12-21; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A laparoscopic group (Active Comparator): group A laparoscopic surgery
  Interventions: Procedure: total mesorectal excision in rectal carcinoma
- Group B (Active Comparator): Group B open surgery
  Interventions: Procedure: total mesorectal excision in rectal carcinoma

INTERVENTIONS:
Procedure: total mesorectal excision in rectal carcinoma — total mesorectal excision laparoscopic versus open technique in management of rectal carcinoma

SUMMARY:
Colorectal cancer is the second leading cause of death in the West, and rectal cancer accounts for about 25% of colon cancers

Low anterior resection has been the mainstay of rectal cancer surgery in low rectal cancer since the 1970s. Although the best efforts of experienced surgeons, The local recurrence rate is 3 to 33% in conventional surgery, while total mesorectal excision (TME) results indicate a recurrence rate of less than 10%

The evolution of the concept of TME which was first revealed by Heald.in 1982 made a major shift in the treatment strategies (Rodriguez-Luna et al,2015). The concept of TME was the most important event in surgery for rectal cancer in the last two decades, because even without a curative approach, the local recurrence decreased to 6 to 12%, and 5-year survival improved by 53-87% TME described clear definitions of distal resection margin (DRM), circumferential resection margin (CRM), and least number of harvested lymph nodes, so oncological outcomes improved, locoregional recurrence and survival rates also influenced .

Laparoscopic total mesorectal excision (LTME) may be associated with less blood loss, earlier recovery, and lower morbidity. Identification of the small nerves and vessels became easiear because of laparoscopic magnified view of pelvis and thus prevents these injuries (Sajid et al, 2019). Also, minimal surgical trauma will reduce the immunologic response and preserves postoperative immunologic defenses. This may lead to low rate of infections as well as low local recurrences and distant metastases in addition to, tissue handling with less manipulation, 'may reduces the spread of cancer cells

TME in obese males with low and anterior rectal tumors is technically challenging especially post neoadjuvant chemoradiotherapy due to distortion of the anatomical planes (Ng et al, 2014). In these patients, it is difficult to obtain a proper view of the dissection plane, in open technique which threatens the integrity of TME and carries the risk of positive margins, which is related to higher rates of local recurrence

LTME is a widely used approach for rectal cancers; although conversion rate varies from 1.2 to 17%, and it is higher if BMI is equal to or more than 30

ELIGIBILITY:
Inclusion Criteria:

* All patients with pathologically confirmed rectal carcinoma involving middle or lower third rectum and operable by MRI and CT scan criteria.
* Both sexes will be included.
* Age: ranging from 20 to 70 years.

Exclusion Criteria:

* Patients with stage IV.
* Recurrent rectal cancers.
* Combined malignancy.
* Patients admitted due to emergency situations (acute large bowel obstruction, abdominal abscess, or rectal perforation and hemorrhage).
* Patients with contraindication for laparoscopic surgery.
* Unfit patients (ASA score > II).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Comparison betewen laparoscopic and open teqnique in resection of rectal carcinoma and the involvement of the resection margin (R1), which is CRM involvement or DRM involvement.after resection. | 1year
  R(resection margin of cancer of rectum) CRM circumferencial margin Or. DRM distal resection margin of cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

REFERENCES:
- [Background] Cecil TD, Sexton R, Moran BJ, Heald RJ. Total mesorectal excision results in low local recurrence rates in lymph node-positive rectal cancer. Dis Colon Rectum. 2004 Jul;47(7):1145-9; discussion 1149-50. doi: 10.1007/s10350-004-0086-6. Epub 2004 Jun 3. PMID 15164243
- [Background] Braga M, Frasson M, Vignali A, Zuliani W, Capretti G, Di Carlo V. Laparoscopic resection in rectal cancer patients: outcome and cost-benefit analysis. Dis Colon Rectum. 2007 Apr;50(4):464-71. doi: 10.1007/s10350-006-0798-5. PMID 17195085
- [Background] Hill GL, Rafique M. Extrafascial excision of the rectum for rectal cancer. Br J Surg. 1998 Jun;85(6):809-12. doi: 10.1046/j.1365-2168.1998.00735.x. PMID 9667714